CLINICAL TRIAL: NCT05588934
Title: A Head-to-Head Comparison of the 2B-Alert Caffeine Optimization Algorithm Versus Standard Caffeine Dosing on Performance During Sleep Deprivation (2B-2)
Brief Title: Caffeine Optimization Versus Standard Caffeine Dosage (2B-2)
Acronym: 2B-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); Biotechnology High Performance Computing Software Applications Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: STUDY00001953
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Sleep Deprivation; Caffeine
Keywords: SLEEP; CAFFEINE
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: There are four different experimental conditions and one control condition that determines the ratio of caffeine gum to placebo gum that is administered to participants.
  1. Standard Caffeine Dose Both Nights (200mg/2 hr. up to 800mg/24 hr.)
  2. Optimized Caffeine Dose Both Nights (0-300mg/2 hr. up to 800mg/24 hr.)
  3. Placebo Dose 1st Night/Standard Caffeine Dose 2nd Night (0mg) / (200mg/2 hr. up to 800mg/24 hr.)
  4. Placebo Dose 1st Night/Optimized Caffeine Dose 2nd Night (0mg) / (0-300mg/2 hr. up to 800mg/24 hr.)
  5. Placebo Dose Both Nights (0mg) Participants will be randomly assigned to 1 of the 5 conditions, so 20% of the study population will be in each condition.
Who Masked: Participant, Investigator
Masking Description: Participants will not have any knowledge of which of the five condition groups they are apart of during or after the study.
  The investigator will not have any knowledge of which of the five condition groups the participant is apart of during or after the study.
  A third party will prepare the caffeine dosing and not participate in the administration to avoid knowledge of what participants are in what categories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo Dose Both Nights (Placebo Comparator): Participants will be administer non-caffeinated, placebo gum during both nights of Phase 2.
  Interventions: Other: Placebo Gum
- Standard Caffeine Dose Both Nights (Active Comparator): Participants will be administer the standard caffeine recommendation (200mg/2 hr. up to 800mg/24 hr.) using caffeinated and non-caffeinated gum during both nights of Phase 2.
  Interventions: Dietary Supplement: Caffeine Gum; Other: Placebo Gum
- Optimized Caffeine Dose Both Nights (Active Comparator): Participants will be administer the optimized caffeine recommendation (0-300mg/2 hr. up to 800mg/24 hr.) potentially using caffeinated and non-caffeinated gum, depending on optimized dosage, during both nights of Phase 2.
  Interventions: Dietary Supplement: Caffeine Gum; Other: Placebo Gum
- Placebo Dose 1st Night/Standard Caffeine Dose 2nd Night (Active Comparator): Participants will be administer non-caffeinated, placebo gum during the first night of Phase 2. Then, participants will be administer the standard caffeine recommendation (200mg/2 hr. up to 800mg/24 hr.) using caffeinated and non-caffeinated gum during the second night of Phase 2.
  Interventions: Dietary Supplement: Caffeine Gum; Other: Placebo Gum
- Placebo Dose 1st Night/Optimized Caffeine Dose 2nd Night (Active Comparator): Participants will be administer non-caffeinated, placebo gum during the first night of Phase 2. Then, participants will be administer the optimized caffeine recommendation (0-300mg/2 hr. up to 800mg/24 hr.) potentially using caffeinated and non-caffeinated gum, depending on optimized dosage, during the second night of Phase 2.
  Interventions: Dietary Supplement: Caffeine Gum; Other: Placebo Gum

INTERVENTIONS:
Dietary Supplement: Caffeine Gum — Commercially available caffeinated gum that contains 100mg of caffeine per piece of gum.
  Other Names: Military Energy Gum
  Arms: Optimized Caffeine Dose Both Nights; Placebo Dose 1st Night/Optimized Caffeine Dose 2nd Night; Placebo Dose 1st Night/Standard Caffeine Dose 2nd Night; Standard Caffeine Dose Both Nights
Other: Placebo Gum — Commercially available non-caffeinated gum.

SUMMARY:
This clinical trial will be a comparison between personalized recommended caffeine dosing regimen versus the standard recommended caffeine dosing regimen for sustaining performance during sleep deprivation and minimizing side effects and subsequent sleep disruption. The questions this study aims to answer are: Whether the personalized caffeine recommendations improve vigilance, sleepiness, and cognition after total sleep deprivation, compared to standard recommendations; Whether the personalized caffeine recommendation better addresses the physical and emotional side effects of total sleep deprivation, compared to standard recommendations; And whether personalized caffeine recommendations aids in better recovery sleep after total sleep deprivation, compared to standard recommendations.

Participants will be asked to:

1. Complete a 13-day at-home portion, wearing an actigraph watch to measure activity and sleep, and complete motor vigilance tests up to six times a day.
2. Complete a 4-day in-lab portion, where participants will have to complete one night of baseline sleep, undergo 62-hours of total sleep deprivation, and then complete one night of recovery sleep.
3. During the in-lab portion of the study, participants will be asked to complete more motor vigilance tests.

Researchers will be comparing the personalized caffeine recommendation group against the standard caffeine recommendation to see if it is better at addressing each of the main questions.

DETAILED DESCRIPTION:
This clinical trial will be examining whether the 2B-Alert Caffeine Optimization algorithm provides greater performance optimization, side effect minimization, and quality of recovery sleep during sleep deprivation compared to the standard published recommendations for caffeine use. The objective of this clinical trial will be to conduct a head-to-head comparison between the 2B-Alert app versus a commonly recommended caffeine dosing regimen for sustaining optimal performance during sleep deprivation and minimizing side effects and subsequent sleep disruption. The specific aims are to: Determine the effectiveness of 2B-Alert versus standard caffeine dosing on psychomotor vigilance, subjective sleepiness, and cognition on single and multiple nights of sleep deprivation; Determine the effectiveness of 2B-Alert versus standard caffeine dosing at mitigating physiological and emotional side effects; Determine the effectiveness of 2B-Alert versus standard caffeine dosing at minimizing disruptions in recovery sleep.

This clinical trial will consist of three phases. Phase 1 includes the enrollment visit where participants will come into the lab, complete baseline personality and mood testing, and be given the actigraph watch and phone with the 2B-Alert app. Then the participant will undergo 13-days of at-home psychomotor vigilance testing and sleep data collection.

Phase 2 begins with the participant arrives at the lab for the 4-day in-lab portion of the study. During this phase the participant will complete a night of baseline sleep using polysomnography to collect sleep data. At the end of baseline sleep, the participant will begin the 62-hour sleep deprivation portion. During the deprivation portion, data will be collected periodically on the participants psychomotor vigilance. After 37-49 hours of continuous sleep deprivation participants will be administered either caffeine gum or placebo gum.

There are four different experimental conditions and one control condition that determines the ratio of caffeine gum to placebo gum that is administered to participants:

1. Standard Caffeine Dose Both Nights (200mg/2 hr. up to 800mg/24 hr.)
2. Optimized Caffeine Dose Both Nights (0-300mg/2 hr. up to 800mg/24 hr.)
3. Placebo Dose 1st Night/Standard Caffeine Dose 2nd Night (0mg) / (200mg/2 hr. up to 800mg/24 hr.)
4. Placebo Dose 1st Night/Optimized Caffeine Dose 2nd Night (0mg) / (0-300mg/2 hr. up to 800mg/24 hr.)
5. Placebo Dose Both Nights (0mg) Participants will be randomly assigned to 1 of the 5 conditions, so 20% of the study population will be in each condition.

After the 62-hour period of total sleep deprivation, participants will complete Phase 3, a night of recovery sleep; During this phase, participants' sleep data will be collected using polysomnography. After the night of recovery sleep participants will remain in the lab for further psychomotor vigilance testing. Once this is complete individuals will be released from the lab and their participation will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 years of age
* Must demonstrate adequate comprehension of the protocol by achieving a score of at least 80% correct on a short multiple-choice quiz

Exclusion Criteria:

* Self-reported habitual nightly sleep amounts outside the target range of approximately 6-9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average)
* Self-reported nighttime bedtimes earlier than approximately 2100 hours on average during weeknights (Sunday through Thursday)
* Self-reported morning wake-up times later than approximately 0900 on average during weekdays (Monday through Friday)
* Self-reported habitual napping (> 3 times per week)
* Self-reported symptoms suggestive of a sleep disorder (to include but not limited to sleep disordered breathing/sleep apnea, narcolepsy, idiopathic hypersomnia, restless leg syndrome, parasomnias, rapid eye movement (REM) behavior disorder, etc.)
* History of a sleep disorder (to include all of the above)
* Any use of prescription or over-the-counter sleep aids during the 6-month period prior to screening indicative of a potential sleep disorder as determined by the examining study physician
* History of neurologic disorder (e.g., seizure disorder, amnesia for any reason, hydrocephalus, multiple sclerosis)
* Self-reported caffeine use > 400 mg per day on average
* Score of 14 or above on the Beck Depression Inventory (BDI)
* Score of 41 or above on the Spielberger Trait Anxiety Inventory (STAI-T)
* Score below 31 or above 69 on the Morningness-Eveningness Questionnaire
* Self-reported regular nicotine use (> 1 cigarette or equivalent per week) within the last 1 year) or positive nicotine/cotinine result during screening visit
* Self-reported heavy alcohol use (≥14 drinks per week or as determined by the examining study physician) or positive saliva alcohol result during screening visit
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction)
* Underlying acute or chronic pulmonary disease requiring daily inhaler use
* Kidney disease or kidney abnormalities
* Liver disease or liver abnormalities
* Self-reported history of psychiatric disorder requiring hospitalization or use of psychiatric medication for any length of time
* Self-reported use of products or drugs that cannot be safely discontinued during in-laboratory phases (determined on a case-by-case basis by the examining study physician)
* Self-reported current use of other illicit drugs (to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana) or positive urine drug screen
* (Females only) positive urine pregnancy result
* (Females only) self-reported or suspected current breast-feeding or collecting breast milk
* Resting blood pressure above 140/90 or resting pulse > 110 beats per minute (if a physician performs a repeat measurement, ~20 minutes after original measure, and it is within range, volunteer will not be excluded)
* BMI ≥ 30 (Obese Class I or greater)
* Clinically significant values (as determined by the reviewing study physician) for any hematology or chemistry parameter
* Inability to read and sign consent
* (Military only) failure to obtain required approved official leave to participate
* Failure to cooperate with requirements of the study, e.g. failure to complete 80% of Smart-Psychomotor Vigilance Tests (PVTs) during Phase 1 (Days 2-13)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean psychomotor vigilance test reaction time | Peak Alertness Window: During each overnight sleep deprivation period from 3:00am to 9:00am
  The mean response time to psychomotor vigilance tests during the Peak Alertness Window.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Arizona Psychiatry Department, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. All data that will be shared from this clinical trial will be shared in summary data sets.

REFERENCES:
- [Background] Kamimori GH, Johnson D, Thorne D, Belenky G. Multiple caffeine doses maintain vigilance during early morning operations. Aviat Space Environ Med. 2005 Nov;76(11):1046-50. PMID 16313140
- [Background] Killgore WD, Kahn-Greene ET, Grugle NL, Killgore DB, Balkin TJ. Sustaining executive functions during sleep deprivation: A comparison of caffeine, dextroamphetamine, and modafinil. Sleep. 2009 Feb;32(2):205-16. doi: 10.1093/sleep/32.2.205. PMID 19238808
- [Background] Killgore WDS, Kamimori GH. Multiple caffeine doses maintain vigilance, attention, complex motor sequence expression, and manual dexterity during 77 hours of total sleep deprivation. Neurobiol Sleep Circadian Rhythms. 2020 May 31;9:100051. doi: 10.1016/j.nbscr.2020.100051. eCollection 2020 Nov. PMID 33364521
- [Background] Liu J, Ramakrishnan S, Laxminarayan S, Balkin TJ, Reifman J. Real-time individualization of the unified model of performance. J Sleep Res. 2017 Dec;26(6):820-831. doi: 10.1111/jsr.12535. Epub 2017 Apr 24. PMID 28436072
- [Background] Ramakrishnan S, Wesensten NJ, Balkin TJ, Reifman J. A Unified Model of Performance: Validation of its Predictions across Different Sleep/Wake Schedules. Sleep. 2016 Jan 1;39(1):249-62. doi: 10.5665/sleep.5358. PMID 26518594
- [Background] Ramakrishnan S, Wesensten NJ, Kamimori GH, Moon JE, Balkin TJ, Reifman J. A Unified Model of Performance for Predicting the Effects of Sleep and Caffeine. Sleep. 2016 Oct 1;39(10):1827-1841. doi: 10.5665/sleep.6164. PMID 27397562
- [Background] Reifman J, Kumar K, Wesensten NJ, Tountas NA, Balkin TJ, Ramakrishnan S. 2B-Alert Web: An Open-Access Tool for Predicting the Effects of Sleep/Wake Schedules and Caffeine Consumption on Neurobehavioral Performance. Sleep. 2016 Dec 1;39(12):2157-2159. doi: 10.5665/sleep.6318. PMID 27634801
- [Background] Vital-Lopez FG, Ramakrishnan S, Doty TJ, Balkin TJ, Reifman J. Caffeine dosing strategies to optimize alertness during sleep loss. J Sleep Res. 2018 Oct;27(5):e12711. doi: 10.1111/jsr.12711. Epub 2018 May 28. PMID 29808510